CLINICAL TRIAL: NCT01191671
Title: Feeding and Sociolinguist Profile in Children
Brief Title: Language and Deglutition in Children
Acronym: LDC
Status: Completed | Type: Observational
Sponsor: Fortaleza University (Other)
Responsible Party: Priscilla Mayara Estrela Barbosa, Fortaleza University
Other Study IDs: PMEB001
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2009-05

CONDITIONS: Child; Development
Keywords: Child Development; Child; Daycare centers; Language
MeSH Terms: conditions — Language

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The first years of life are considered essential to child development, as there is greater brain growth and formation of more neural connections. Therefore, the stimulation of children in various fields of development becomes relevant to the acquisition of knowledge and skills.

DETAILED DESCRIPTION:
Child development, food and language, particularly in young children in different socioeconomic and cultural, as this is the basis for the growth conditions, socialization and learning.

ELIGIBILITY:
Inclusion Criteria:

* children aged one to three years of chronological age, of both genders, enrolled full-time, ie more than six hours in childcare elected for search

Exclusion Criteria:

* children with minor changes or deviations in child development, who did at least one major meal (lunch or dinner) in the nursery, or other educational institution attended, in addition

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 89 children, 41 children in public kindergarten and 48 children in daycare facilities.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla ME Barbosa, Graduate, Principal Investigator — University of Fortaleza
Locations (1):
- University of Fortaleza, Fortaleza, Ceará, Brazil